CLINICAL TRIAL: NCT04710641
Title: An Open Label, Randomised Phase 2 Study to Evaluate the Safety and Efficacy of MTL-CEBPA Administered in Combination With Sorafenib or Sorafenib Alone in TKI naïve Participants With Previously Treated Advanced Hepatocellular Carcinoma (HCC) and Hepatitis B or Hepatitis C Virus (OUTREACH2)
Brief Title: Radomised Phase II Study of MTL-CEBPA Plus Sorafenib or Sorafenib Alone
Acronym: OUTREACH2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mina Alpha Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNA-3521-014-RNDZ
Record Dates: First submitted 2021-01-07; First posted 2021-01-15 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma; Hepatitis B; Hepatitis C
Keywords: saRNA; MTL-CEBPA; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B; Hepatitis C | interventions — Sorafenib

STUDY DESIGN:
Intervention Model Description: Participants will be randomised 2:1 to receive either both the experimental drug, MTL-CEBPA, and sorafenib tablets or sorafenib tablets alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MTL-CEBPA in combination with sorafenib (Experimental): Intravenous infusion of MTL-CEBPA 130mg/m2 given once every 3 weeks. Oral sorafenib 400mg twice a day will commence C1D8.
  Interventions: Drug: MTL-CEBPA; Drug: Sorafenib
- Sorafenib alone (Active Comparator): Oral sorafenib 400mg twice a day commencing Day1
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: MTL-CEBPA — Administered once every 3 weeks on Day 1 of each 3 week cycle.
  Arms: MTL-CEBPA in combination with sorafenib
Drug: Sorafenib — Oral adminstration twice a day
  Other Names: Nexavar

SUMMARY:
This is a Phase II study in patients with advanced liver cancer (hepatocellular carcinoma) as a result of hepatitis B and/or C infection. Participants will be dosed with either MTL-CEBPA (an experimental treatment) and sorafenib or sorafenib alone. The MTL-CEBPA is administered once every 3 weeks via intravenous infusion. Sorafenib is taken orally from Day 8 for the combination group or Day 1 for the sorafenib alone group at a dose of 400 mg twice a day. Participants will receive 3 week cycles of treatment until disease progression, unacceptable toxicity, withdrawal of consent or death occurs. The combination of MTL-CEBA and sorafenib combination of treatment was tested in a previous Phase I study (OUTREACH) which showed anti-tumour activity along with a good safety and toxicity profile.

DETAILED DESCRIPTION:
After a participant has signed the consent form to confirm they wish to participate in the study a number of assessments (screening) will be completed to determine whether they are suitable to be enrolled in the study. Prior to the the first dose of experimental drug (MTL-CEBPA) a 2:1 randomisation programme will allocate to which arm the person will be allocated. For participants allocated to the combination treatment arm, MTL-CEBPA will be given via infusion on the first day (Cycle 1 Day 1) of the study. It will subsequently be administered every 21 days. Sorafenib tablets (a drug which is already used to treat liver cancer) will be started on the eighth day of the study and taken daily whilst the participant is in the study. If the participant is tolerating the combination of drugs and there is no evidence that the cancer is advancing they will continue to receive cycles (21 days in length) of treatment. For participants allocated to the single treatment arm, sorafenib tablets will be started on Day 1. All participants will have contrast-enhanced CT scans of the chest, abdomen and pelvis at the beginning of the study and then every 8 weeks whilst in the study. Assessments will be completed throughout the study to ensure the combination of drugs is safe. These will include recording any adverse events (untoward medical occurrences), vital signs (such as blood pressure, pulse, body temperature, and breathing rates), ECG, and completing blood tests. Blood samples, analysed in both local (hospital/clinic site) and central laboratories (ie, facilities independent of hospital/clinic labs) will be taken throughout the study. The maximum amount of blood taken in any 28-day treatment cycle is approximately 182 mL. A patient questionnaire will be used to assess changes in health-related quality of life for participants. The questionnaire will be used for all participants in the study and will be completed every 3 weeks. All participants will be offered an optional liver tumour biopsy prior to being administered study treatment and again if clinically feasible during treatment.

ELIGIBILITY:
1.Written informed consent obtained prior to any specific trial-related procedure.

2.Male or female 18 years or older. 3.Histologically confirmed advanced HCC with cirrhosis in a participant with a history of hepatitis B and/or C. Participants with past or ongoing HCV infection will be eligible for the study. Participants must have completed their treatment at least 1 month prior to starting study intervention and their HCV viral load below the limit of quantification. Participants who are HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution will be eligible. Participants with past or controlled ongoing hepatitis B will be eligible as long as their HBV viral load is less than 500 IU/mL prior to first dose of study drug. Participants on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study intervention.

4.Child-Pugh classification A. 5.Unsuitable for liver tumour resection and/or refractory to loco regional therapy.

6.Not eligible for liver transplantation. 7.Had progression or recurrence of HCC following previous treatment with atezolizumab in combination with bevacizumab. Participants with progression or recurrence of HCC on non-atezolizumab anti-PD-1/PD-L1 inhibitors and non-bevacizumab anti-VEGF agent in combination or as any as single agents, and no prior treatment with atezolizumab and bevacizumab, are eligible.

8.Naïve to tyrosine kinase inhibitors, including sorafenib, regorafenib, cabozantinib, and lenvatinib.

9.Participants with BCLC stage C disease. BCLC Stage B will be allowed if not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach (Appendix B).

10.Eastern Cooperative Oncology Group performance status of 0 or 1. 11.Has the ability to swallow and retain oral medication. 12.Life expectancy greater than 3 months at time of recruitment. 13.At least one measurable liver lesion (RECIST v1.1) assessed by the investigator.

14.Platelet count >70 x109/L. 15.Serum albumin ≥28g/L. 16.Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 x the upper limit of normal (ULN).

17.Bilirubin ≤50 μmol /L. 18.White Blood Cell (WBC) ≥2.0 x 109/L. 19.Absolute neutrophil count ≥1.5 x 109/L. 20.Haemoglobin ≥9.0 g/dL. 21.International Normalized Ratio (INR) <1.5. 22.Calculated creatinine clearance ≥50 mL/min (Cockcroft & Gault). 23.AEs due to prior therapy must have resolved to Grade ≤1 (except alopecia or endocrinopathies that are adequately managed through hormone replacement treatment).

24.Negative blood pregnancy test for women of childbearing potential (within 10 days prior to first drug administration). Note: a woman is considered of child-bearing potential following menarche and until becomingpost-menopausal unless permanently sterile. Permanent methods of sterilisation include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A post-menopausal state is defined as no menses for 12 months without an alternative medical cause.https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf(see additional information / requirements in Section 5.1.) 25.Female participants of childbearing potential must use highly effective* contraceptive measures adequate to prevent a new pregnancy for the duration of the study treatment with MTL-CEBPA and sorafenib and, in addition, for at least six months after the last dose of MTL-CEBPA and six months beyond the last dose of sorafenib, as recommended in sorafenib's U.S. Package Insert (USPI). For women with reproductive potential who use a hormonal method of contraception, concurrent use of a second (barrier) method is recommended. * Highly effective methods of birth control are defined as those that result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly (e.g. implants, injectables, oral contraceptives, some intrauterine devices, bilateral tubal occlusion, true sexual abstinence in line with the preferred and usual lifestyle of the participant, or vasectomised partner). (See additional information / requirements https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_ HMA_CTFG_Contraception.pdf) 26.Male participants with partners of child-bearing potential must use highly effective contraception and are required to use barrier contraception plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least three months after the last dose of MTL-CEBPA. Male participants will also be advised to abstain from sexual intercourse with pregnant or lactating women, or to use condoms. Male participants with partners of child-bearing potential must use highly effective contraception during treatment with sorafenib and for 3 months beyond the last dose of sorafenib, as recommended in sorafenib's USPI.

27.Abstinence is only acceptable if it is line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to IMP, and withdrawal are not acceptable methods of contraception.

28.Able to comply with all the requirements of the protocol. Exclusion Criteria Participants should not enter the study if any of the following exclusion criteria are fulfilled.

1. Child-Pugh classification B and C.
2. Participants without a history of hepatitis B and/or hepatitis C.
3. Participants with fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtype HCC.
4. Participants with no prior therapy who are eligible for first-line treatment with atezolizumab in combination with bevacizumab.
5. Participants who received investigational drug(s) within the last 30 days prior to study treatment initiation.
6. Participants with clinically significant ascites.
7. Any episode of bleeding from oesophageal varices or other uncontrolled bleeding including clinically meaningful epistaxis within the last 3 months prior to study treatment initiation.
8. Clinically diagnosed hepatic encephalopathy in the last 6 months unresponsive to therapy.
9. Participants with a history of gastrointestinal haemorrhage or perforation.
10. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated such metastases may participate provided they are radiologically stable for at least 4 weeks by repeat imaging performed during study screening, clinically stable and without requirement of steroid treatment for at least 28 days prior to first dose of study intervention. MRI brain scan are required for all participants with stable brain metastases at screening (CT scan will be allowed if MRI is contraindicated).
11. Participants administered with serum albumin within the last 7 days prior to the first study treatment administration.
12. Known infection with human immunodeficiency virus (HIV) with CD4+ T-cell counts <350cells/μL or with a history of AIDS-defining opportunistic infection. No HIV testing is required unless mandated by local health authority.
13. Received a live vaccine within 30 days prior to the first dose of study treatment.Live vaccines include, but are not limited to: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccinesfor injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
14. Known other malignancy that is progressing or has required active treatment in the last 5years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death such as early-stage cancers treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy.
15. Participants presenting with a baseline prolongation of QT/QTc interval defined as repeated demonstration of a QTc interval ≥450ms (males) and ≥460ms (females) using Fridericia's correction formula.
16. Participants with a screening diastolic blood pressure >90 mm Hg.
17. Clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability. Note: Medically controlled arrhythmia would be permitted.
18. Major surgery within the last 30 days prior to study treatment initiation. If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
19. Participants with a history of organ transplantation.
20. Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy.
21. Participants with sepsis, ineffective biliary drainage with or without cholangitis, obstructive jaundice, or encephalopathy at screening visit or within the last 2 weeks prior to study treatment initiation.
22. Evidence of spontaneous bacterial peritonitis or renal failure, or allergic reaction at screening visit or within the last two weeks prior to study treatment initiation, whichever is earlier.
23. Pregnant or lactating women.
24. Known hypersensitivity to the active substance or to any of the excipients of both MTL-CEBPA and sorafenib.
25. History or evidence of any other condition or therapy, including a known psychiatric or substance abuse disorder that, in the judgment of the investigator, may interfere with the study conduct or confound the results, pose a risk to the participant, is not in their best interest to take part, or may affect their ability to follow the protocol specific procedures for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From baseline CT scan until end of documented progression or date of death from any cause assessed up o 100 weeks
  Change from baseline CT scan using blinded central review of Response Evaluation Criteria in Solid Tumours v.1.1 and compare between the two arms

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL) questionnaires | From first cycle of treatment to end of study approximately one year
  To compare the health-related quality of life (HRQoL) of MTL-CEBPA in combination with sorafenib compared to sorafenib alone as assessed by EORTC-QLQ-C30 plus EORTC-QLQ-HCC18 QOL questionnaires.
Overall survival (OS) | From first dose of MTL-CEBPA and sorafenib or sorafenib alone to end of treatment
  To compare overall survival (OS) between the two arms using statistical analysis
Adverse events | From first dose of MTL-CEBPA and sorafenib or sorafenib alone to end of treatment
  Compare the incidence of AEs/serious AEs (SAE) graded according to toxicity criteria (CTCAE v5.0 between the two arms

CONTACTS AND LOCATIONS:
Locations (2):
- City of Hope, Duarte, California, United States
- National University Hospital Singapore, Singapore, Singapore

REFERENCES:
- See also: Sponsor website — http://www.minatx.com